CLINICAL TRIAL: NCT01416025
Title: A Prospective, Randomized Trial Comparing the Efficacy and Safety of Voriconazole Administered With Therapeutic Drug Monitoring vs. Standard Dosing
Brief Title: A Trial Comparing Efficacy and Safety of Voriconazole Administered With Therapeutic Drug Monitoring vs. Standard Dosing
Acronym: VoriTDM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Kieren Marr, Professor of Medicine and Oncology, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00041916
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Fungal Infection
Keywords: Voriconazole; Therapeutic drug monitoring; Hematopoietic stem cell transplant; Hematologic malignancy; Invasive mould infection
MeSH Terms: conditions — Mycoses; Hematologic Neoplasms | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prospective TDM Arm (Experimental): Voriconazole dose will be adjusted based on per protocol obtained TDM levels
  Interventions: Drug: Prospective TDM Arm
- Standard dosing (No Intervention): Standard doses of voriconazole will be used

INTERVENTIONS:
Drug: Prospective TDM Arm — Voriconazole dose will be adjusted based on per protocol obtained TDM levels
  Other Names: VFEND
  Arms: Prospective TDM Arm

SUMMARY:
This is a prospective, multicenter, randomized trial to study therapeutic drug monitoring (TDM) of voriconazole among patients with an invasive mould infection (IMI). The primary objective of this study will be to assess the effect of prospective voriconazole TDM on the composite of adverse events (AE) and clinical response.

DETAILED DESCRIPTION:
This is a prospective study of patients who receive voriconazole as treatment for an IMI (proven, probable, and possible by the EORTC/MSG definitions), other than zygomycosis. Patients will be randomized to receive either standard dosing or dosing based on TDM, stratified by whether initial voriconazole therapy is PO or IV. Assessment of outcomes will be made 42 days after start of voriconazole. An additional follow up for safety reporting will be performed 4weeks after completion of voriconazole

The patients will be randomized to:

* Prospective TDM: voriconazole dose will be adjusted based on per protocol obtained TDM levels, and
* Standard dosing: standard doses of voriconazole will be used.

In the prospective TDM arm, voriconazole TDM will be performed in real time at each site and results will be reported to treating physicians for dose adjustment. All efforts will be taken to obtain results within 24 hours of blood sample collection. In the standard dosing arm, blood samples will be collected, stored, and batched for voriconazole levels to be tested retrospectively. Voriconazole plasma levels will be measured by validated high performance liquid chromatography (HPLC) assays as detailed. Voriconazole trough levels will be performed on Day Baseline/Screening, 5, 14, 28, and 42.

Voriconazole peak level will be measured on Day 5. Trough voriconazole levels will be obtained in case of an event, defined as suspected drug-associated toxicity and/or clinical failure.

Assessment of AEs for all patients will be monitored during the study and response to treatment will be assessed. The composite of overall AE/clinical failure will be assessed on day 42.

ELIGIBILITY:
Inclusion Criteria:

* Indication for voriconazole administration: proven, probable, or possible IMI, excluding zygomycosis (based on the revised EORTC/MSG consensus definitions) [De Pauw, Clin Infect Dis. 2008; 46:1813].
* Male or female ≥12 years of age.
* Evidence of a personally signed and dated informed consent document in accordance with local regulatory and legal requirements indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Known history of allergy, hypersensitivity or serious reaction to azole antifungals.
* Patients with aspergilloma or allergic bronchopulmonary aspergillosis (ABPA).
* Patients with chronic invasive aspergillosis with duration of symptoms or radiological finding for more than 4 weeks prior to study entry.
* Patients who are receiving and cannot discontinue the following drugs at least 24 hours prior to randomization: terfenadine, pimozide or quinidine (because of the possibility of QT prolongation), St John's wort preparation.
* Patients receiving any of the following medications: sirolimus, rifampin, rifabutin, carbamazepine, long acting barbiturates (e.g., phenobarbital, mephobarbital), ritonavir, efavirenz, or ergot alkaloids (e.g., ergotamine, dihydroergotamine).
* Receipt of more than 5 days of voriconazole as treatment prior to enrollment.
* Receipt of 7 days or more of systemic antifungal treatment for the current episode of IMI.
* Severe liver dysfunction (defined as total bilirubin, AST, ALT, or alkaline phosphatase >5x upper limit of normal). Local laboratory results may be used to qualify individuals for enrollment.
* Patients with any condition which, in the opinion of the investigator, could affect patient safety, preclude evaluation of response, or make it unlikely that the proposed course of therapy can be completed.
* Patients who have already participated in this trial within the last 30 days.
* Patients with a high likelihood of death due to factors unrelated to IA (e.g., due to relapsed malignancy, severe GVHD, other underlying diseases, etc.) within 30 days following planned enrollment (investigator's discretion).
* Patients that weigh <45 and >120 kg, respectively, upon enrollment. If patients' weight is beyond those limits upon serial assessments during the study period, the study monitor should be contacted and decisions to keep or withdraw subject from the study will be made.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kieren Marr, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective TDM Arm | Standard Dosing
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective TDM Arm | Standard Dosing | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Full Range); unit: years] | 63.4 [49 to 83] | 59.1 [28 to 84] | 62.5 [28 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Failure
Description: The primary endpoint of the study will be a binary outcome, called Failure, defined as one of the following: measured at 42 days from initiation of drug administration:
  1. Progression of underlying infection (clinical failure)
  2. Death
  3. Development of a voriconazole-associated SAE: LFTs, Rash, Visual disturbance, Neurologic abnormality (e.g: hallucinations)
Time Frame: 42 days
Measure: Number; unit: participants
Arm/Group | Prospective TDM Arm | Standard Dosing
Number analyzed (Participants) | 14 | 15
participants | 1 | 5

ADVERSE EVENTS:
Arm/Group | Prospective TDM Arm | Standard Dosing
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/15
Other Adverse Events (participants affected / at risk) | 3/14 | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospective TDM Arm (N=14) | Standard Dosing (N=15)
hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prospective TDM Arm (N=14) | Standard Dosing (N=15)
Stop voriconazole (Psychiatric disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No